CLINICAL TRIAL: NCT02983110
Title: Does Sex Hormone Therapy Decrease Nucleos(t)Ide Reverse Transcriptase Inhibitors (NRTI) Active Metabolite Formation in Mucosal Tissues?
Brief Title: Sex Hormone Therapy and Mucosal Tissues
Acronym: SHAMT
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 16-2122
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Hiv
Keywords: Hormones, Transgender
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Proctoscopy; Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort B: Group B will be HIV Infected post-menopausal women who are not receiving hormonal therapy to provide tissue, blood, and cells
  Interventions: Procedure: Anoscopy with Rectal Tissue Sampling; Procedure: Phlebotomy; Procedure: Female Genital Tract Sampling
- Cohort C: Group C will be HIV infected transgendered women receiving hormone therapy to provide tissue and blood
  Interventions: Procedure: Anoscopy with Rectal Tissue Sampling; Procedure: Phlebotomy
- Cohort E: Group E will be HIV infected men
  Interventions: Procedure: Anoscopy with Rectal Tissue Sampling; Procedure: Phlebotomy

INTERVENTIONS:
Procedure: Anoscopy with Rectal Tissue Sampling — All subjects will provide 10 pieces of rectal tissue
Procedure: Phlebotomy — • Procedure: Blood plasma/serum collection Approximately 17 mL of blood will be taken from each subject just prior to tissue sampling.
Procedure: Female Genital Tract Sampling — Cohorts B only will have cervical cells, cervical tissue, and vaginal tissue collected
  Groups: Cohort B

SUMMARY:
The purpose of this research study is to better understand how sex hormone therapy that is used to treat women for menopausal symptoms, men with low testosterone, or as hormone therapy for transgender women, affects a class of medications called NRTIs (nucleoside reverse transcriptase inhibitors) used to treat and prevent HIV infection. The two most commonly used NRTIs are tenofovir and emtricitabine, which are the components of the drug Truvada and also included in the combination products Atripla, Complera, and Stribild. The medication's ability to work effectively may be altered when someone is also taking sex hormone therapy.

In order to determine this effect, samples will be collected from some parts of the body where HIV makes copies. These samples will be measured for the levels of HIV medication, HIV virus and sex hormones that are present. The samples that will be looked at in this study include blood, cells from the vagina, semen, and tissue biopsies from the female genital tract and rectum.

DETAILED DESCRIPTION:
Study Design:

This is an observational study of tenofovir/emtricitabine (TFV/FTC) concentrations in the genital and lower gastrointestinal tracts. Participants will be selected on the basis of receiving TFV/FTC as part of their ongoing HIV care. After participant education, informed consent, and screening for study eligibility, participants will be evaluated at baseline. All samples will be collected over the course of an outpatient sampling visit.

Study Sampling:

1. A blood sample will be collected to measure the concentration of TFV/FTC in the blood plasma, the concentration of TFV/FTC active metabolite concentrations (TFVdp/FTCtp) in the PBMCs, and the concentration of sex hormones in the blood stream.
2. Vaginal and cervical tissue will be collected (for cisgender women) to measure for concentrations of TFVdp/FTCtp, HIV RNA, and estrogen/progesterone.
3. Rectal tissue samples will be collected to measure for concentrations of TFVdp/FTCtp, HIV RNA, estrogen/progesterone (for cisgender and transgender women), and testosterone (for cisgender men).
4. A semen sample will be collected (for cisgender men) to measure the concentrations of TFV/FTC, HIV RNA and testosterone.

Pharmacokinetic Analysis:

All blood, cervical, vaginal, semen and rectal tissue samples will be analyzed by the Clinical Pharmacology and Analytical Chemistry Laboratory (CPAC) at the UNC School of Pharmacy. TFV/FTC will be measured in blood and seminal plasma and TFVdp/FTCtp will be measured in PBMCs, SMCs using validated LC-MS/MS methods. HIV RNA will be measured in blood and seminal plasma using the Abbott Real Time HIV-1 quantitative assay. HIV RNA within the cervical and seminal cells and rectal tissues will be measured using an established Droplet Digital PCR method. Estradiol and progesterone will be measured in serum using validated florescent immunoassays.

ELIGIBILITY:
Inclusion Criteria:

-

All subjects eligible to enroll must meet the following inclusion criteria, regardless of cohort:

* HIV-positive adults aged 18-65, inclusive on the date of screening, clinically healthy, with an intact gastrointestinal tract. Any screening test may be repeated once in the screening window to confirm or verify eligibility.
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all the pertinent details of the study.
* Willing and able to comply with scheduled visits, treatment plan laboratory tests, and other trial procedures
* Subjects must not be actively involved in the conception process, currently pregnant/lactating/ or in the immediate post-partum period.
* Subjects must be willing to abstain from all sexual activity, and all intravaginal and intrarectal products for at least 72 hours prior to the sampling day, until seven days later
* HIV RNA viral load undetectable (<50 copies/mL or less per institution) within at least the previous six months prior to screening. Repeat HIV RNA Viral load testing may be conducted at screening, if indicated.

  -->80% adherent to their antiretroviral regimen per self-report, and a compliant diary card 5 days before intensive sampling
* Actively adherent to an antiretroviral regimen containing both tenofovir (TDF) and emtracitabine (FTC) for >1 month (if switched from previous regimen) or >3 months (if previously antiretroviral naive) as part of their standard clinic care
* Negative, or treated, sexually transmitted infections at screening including syphilis, gonorrhea, chlamydia, and trichomoniasis
* All subjects must have an estimated calculated creatinine clearance of (eCcr) at least 60mL/min by the Cockcroft-Gault formula
* No clinical or surgical abnormalities (i.e. hysterectomy) that would preclude sample collection
* Hemoglobin Grade 2 or lower, with no clinical significant medical issues that would preclude blood sampling
* Coagulation testing Grade 2 or lower, with no clinically significant medical issues that would preclude tissue sampling

Exclusion Criteria:

* Age outside of desired range
* Subject is HIV negative
* Impaired renal function, as documented with a creatinine clearance <60mL/min with the Cockcroft-Gault equation
* Receiving an antiretorivral regimen that does not include TDF/FTC, or adherent to a TDF/FTC regimen less than one month, or patient is unlikely to remain on this regimen during the sampling period
* Less than 80% adherence to anti-retroviral medications, and more than 3 missed doses in the month preceding enrollment
* Subject is not able or willing to follow the diet and lifestyle guidelines necessary for the study period
* Active, untreated, sexually transmitted infection, including syphilis, gonorrhea, chlamydia or trichomoniasis or symptomatic bacterial vaginosis
* Clinical, laboratory, or surgical abnormalities that would preclude sample collection (for example but not limited to: hysterectomy)
* Subjects actively involved in the conception process, currently pregnant or lactating, or immediately post-partum

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will consist of 20 HIV positive men and women between 18-65 years of age (inclusive) with an intact gastrointestinal tract, uterus/cervix (if cisgender women), and male genital tract (if cisgender man) who are available to complete all study procedures at UNC.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Quantification of tenofovir/emtricitabine active metabolite (TFVdp/FTCtp) concentrations in ectocervical/vaginal (cisgender women) and rectal (all cohorts) tissue biopsies by LC-MS/MS. | Samples collected within 24 hours post-dose
  (TFVdp/FTCtp)
Quantification of tenofovir/emtricitabine active metabolite (TFVdp/FTCtp) concentrations in PBMCs (all cohorts) and seminal mononuclear cells (cisgender men). | Samples collected within 24 hours post-dose
  PBMC concentrations

SECONDARY OUTCOMES:
Quantification of HIV RNA concentrations | Samples collected within 24 hours post-dose
  in the female tract cells (cisgender women), seminal cells (cisgender men) and rectal tissue (all cohorts) by Droplet Digital PCR method and within seminal (cisgender men) and blood plasma (all cohorts) by Abbott R
Quantification of estradiol/progesterone (cisgender and transgender women) and testosterone (cisgender men) concentrations in blood serum. | Samples collected within 24 hours post-dose
  hormone concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Mackenzie Cottrell, PharmD, Principal Investigator — UNC Chapel Hill
Locations (1):
- Clinical and Translational Research Center, UNC Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cottrell ML, Yang KH, Prince HM, Sykes C, White N, Malone S, Dellon ES, Madanick RD, Shaheen NJ, Hudgens MG, Wulff J, Patterson KB, Nelson JA, Kashuba AD. A Translational Pharmacology Approach to Predicting Outcomes of Preexposure Prophylaxis Against HIV in Men and Women Using Tenofovir Disoproxil Fumarate With or Without Emtricitabine. J Infect Dis. 2016 Jul 1;214(1):55-64. doi: 10.1093/infdis/jiw077. Epub 2016 Feb 24. PMID 26917574
- [Background] Nicol MR, Fedoriw Y, Mathews M, Prince HM, Patterson KB, Geller E, Mollan K, Mathews S, Kroetz DL, Kashuba AD. Expression of six drug transporters in vaginal, cervical, and colorectal tissues: Implications for drug disposition in HIV prevention. J Clin Pharmacol. 2014 May;54(5):574-83. doi: 10.1002/jcph.248. Epub 2014 Jan 2. PMID 24343710
- [Background] Cottrell ML, Prince HM, Allmon A, Mollan KR, Hudgens MG, Sykes C, White N, Malone S, Dellon ES, Madanick RD, Shaheen NJ, Patterson KB, Kashuba AD. Cervicovaginal and Rectal Fluid as a Surrogate Marker of Antiretroviral Tissue Concentration: Implications for Clinical Trial Design. J Acquir Immune Defic Syndr. 2016 Aug 15;72(5):498-506. doi: 10.1097/QAI.0000000000000996. PMID 26999532
- [Derived] Cottrell ML, Prince HMA, Schauer AP, Sykes C, Maffuid K, Poliseno A, Chun TW, Huiting E, Stanczyk FZ, Peery AF, Dellon ES, Adams JL, Gay C, Kashuba ADM. Decreased Tenofovir Diphosphate Concentrations in a Transgender Female Cohort: Implications for Human Immunodeficiency Virus Preexposure Prophylaxis. Clin Infect Dis. 2019 Nov 27;69(12):2201-2204. doi: 10.1093/cid/ciz290. PMID 30963179